CLINICAL TRIAL: NCT01223404
Title: Nicotinic Modulation of the Default Network of Resting Brain Function
Brief Title: Nicotinic Modulation of the Default Network
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Britta Hahn, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HP-00042696; R21DA027894 (NIH)
Record Dates: First submitted 2010-10-13; First posted 2010-10-19 (Estimated); Results first posted 2018-01-25 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Magnetic Resonance Imaging; Cognition; Nicotine; Mecamylamine
Keywords: nicotine; mecamylamine; attention; default network; fMRI
MeSH Terms: interventions — Nicotine; Mecamylamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the statistician performing the randomization and the pharmacist dispensing the drugs were aware which drug was given on which day.
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo, Nicotine, Mecamylamine (Experimental): Participants undergo 3 test sessions:
  In the first session ("placebo"), a placebo patch and a placebo capsule is administered.
  In the second session ("nicotine"), a nicotine patch (7 mg/24 hrs) and a placebo capsule is administered.
  In the third session ("mecamylamine"), a placebo patch and a mecamylamine capsule is administered.
  Interventions: Drug: Placebo; Drug: Nicotine; Drug: Mecamylamine
- Nicotine, Placebo, Mecamylamine (Experimental): Participants undergo 3 test sessions:
  In the first session ("nicotine"), a nicotine patch and a placebo capsule is administered.
  In the second session ("placebo"), a placebo patch (7 mg/24 hrs) and a placebo capsule is administered.
  In the third session ("mecamylamine"), a placebo patch and a mecamylamine capsule is administered.
  Interventions: Drug: Placebo; Drug: Nicotine; Drug: Mecamylamine
- Placebo, Mecamylamine, Nicotine (Experimental): Participants undergo 3 test sessions:
  In the first session ("placebo"), a placebo patch and a placebo capsule is administered.
  In the second session ("mecamylamine"), a placebo patch (7 mg/24 hrs) and a mecamylamine capsule is administered.
  In the third session ("nicotine"), a nicotine patch and a placebo capsule is administered.
  Interventions: Drug: Placebo; Drug: Nicotine; Drug: Mecamylamine
- Nicotine, Mecamylamine, Placebo (Experimental): Participants undergo 3 test sessions:
  In the first session ("nicotine"), a nicotine patch and a placebo capsule is administered.
  In the second session ("mecamylamine"), a placebo patch (7 mg/24 hrs) and a mecamylamine capsule is administered.
  In the third session ("placebo"), a placebo patch and a placebo capsule is administered.
  Interventions: Drug: Placebo; Drug: Nicotine; Drug: Mecamylamine
- Mecamylamine, Placebo, Nicotine (Experimental): Participants undergo 3 test sessions:
  In the first session ("mecamylamine"), a placebo patch and a mecamylamine capsule is administered.
  In the second session ("placebo"), a placebo patch (7 mg/24 hrs) and a placebo capsule is administered.
  In the third session ("nicotine"), a nicotine patch and a placebo capsule is administered.
  Interventions: Drug: Placebo; Drug: Nicotine; Drug: Mecamylamine
- Mecamylamine, Nicotine, Placebo (Experimental): Participants undergo 3 test sessions:
  In the first session ("mecamylamine"), a placebo patch and a mecamylamine capsule is administered.
  In the second session ("nicotine"), a nicotine patch (7 mg/24 hrs) and a placebo capsule is administered.
  In the third session ("placebo"), a placebo patch and a placebo capsule is administered.
  Interventions: Drug: Placebo; Drug: Nicotine; Drug: Mecamylamine

INTERVENTIONS:
Drug: Placebo — Participants are administered a placebo patch and a placebo capsule
Drug: Nicotine — Participants are administered a nicotine patch (7 mg/24 hrs) and a placebo capsule
  Other Names: Nicotine CQ
Drug: Mecamylamine — Participants are administered a placebo patch and a capsule containing 7.5 mg of mecamylamine

SUMMARY:
Many disorders where attentional problems are a hallmark, such as Alzheimer's disease and schizophrenia, display abnormal regulation of the so-called default network of resting brain function that maintains internally directed thought when the mind is free to wander. There is indication that nicotine may improve attention by aiding the deactivation of the default network, and this mechanism may be of therapeutic benefit for the above disease states. The current project aims at providing a proof of concept by demonstrating that nicotinic drugs modulate default network function. The nicotinic agonist nicotine is hypothesized to improve attention by facilitating the down-regulation of default network activity, and the nicotinic antagonist mecamylamine is hypothesized to impair attention by impeding the down-regulation of default network activity during attentional task performance.

DETAILED DESCRIPTION:
This study only enrolls healthy non-smokers. Participants perform attention tasks while undergoing functional Magnetic Resonance Imaging on three separate days. Across the three days, three difference conditions are tested in a double-blind manner, in randomized order. In all test sessions, participants receive a skin patch and swallow a capsule. In one session, both are a placebo. In another, the patch is a low-dose nicotine patch, and the capsule is a placebo. In another session, the patch is a placebo and the capsule contains a low dose of mecamylamine.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 through 50.
* Did not consume cigarettes, cigarillos, cigars, or other tobacco or nicotine-containing products more than 20 times in lifetime, and did not use any nicotine-containing product at all within the last two years.
* Normal or corrected to normal vision (at least 20/80).

Exclusion Criteria:

* Presence of metal objects in the body, implanted electronic devices, or any other counter indication for MRI.
* Claustrophobia.
* Major psychiatric disorders including mood, anxiety or psychotic disorders.
* Cardiovascular or cerebrovascular disease, such as history of myocardial infarction, heart failure, angina, stroke, severe arrhythmias, or EKG abnormalities.
* Kidney or liver disease.
* Hypertension (resting systolic BP above 140 or diastolic above 85 mm Hg).
* Hypotension (resting systolic BP below 95 or diastolic below 60).
* Use of any prescription or over-the-counter drug other than supplements and birth control.
* History of or current neurological illnesses, such as stroke, seizures, dementia or organic brain syndrome.
* Learning disability, attention deficit disorder, or any other condition that impedes memory and attention.
* Glaucoma, organic pyloric stenosis, uremia or renal insufficiency.
* Prostatic hypertrophy, bladder neck obstruction or urethral stricture.
* Left-handed or ambidextrous.
* Pregnant as determined by urine test, or breast-feeding.
* History or current diagnosis of drug or alcohol abuse or dependence.
* IQ < 85 as estimated by the WASI vocabulary subtest.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Britta Hahn, Ph.D., Principal Investigator — University of Maryland, College Park
Locations (2):
- United States (2):
  - National Institute on Drug Abuse, Intramural Research Program, Baltimore, Maryland
  - Maryland Psychiatric Research Center, Baltimore, Maryland

REFERENCES:
- [Background] Hahn B, Ross TJ, Yang Y, Kim I, Huestis MA, Stein EA. Nicotine enhances visuospatial attention by deactivating areas of the resting brain default network. J Neurosci. 2007 Mar 28;27(13):3477-89. doi: 10.1523/JNEUROSCI.5129-06.2007. PMID 17392464

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo, Nicotine, Mecamylamine: First session: Placebo patch and placebo capsule (filler: methylcellulose) Second session: Nicotine patch and Placebo capsule (filler: methylcellulose) Third session: Placebo patch and Mecamylamine capsule
- Nicotine, Placebo, Mecamylamine: First session: Nicotine patch and placebo capsule (filler: methylcellulose) Second session: Placebo patch and Placebo capsule (filler: methylcellulose) Third session: Placebo patch and Mecamylamine capsule
- Placebo, Mecamylamine, Nicotine: First session: Placebo patch and Placebo capsule (filler: methylcellulose) Second session: Placebo patch and Mecamylamine capsule Third session: Nicotine patch and Placebo capsule (filler: methylcellulose)
- Nicotine, Mecamylamine, Placebo: First session: Nicotine patch and placebo capsule (filler: methylcellulose) Second session: Placebo patch and Mecamylamine capsule Third session: Placebo patch and Placebo capsule (filler: methylcellulose)
- Mecamylamine, Placebo, Nicotine: First session: Placebo patch and Mecamylamine capsule Second session: Placebo patch and Placebo capsule (filler: methylcellulose) Third session: Nicotine patch and Placebo capsule (filler: methylcellulose)
- Mecamylamine, Nicotine, Placebo: First session: Placebo patch and Mecamylamine capsule Second session: Nicotine patch and Placebo capsule (filler: methylcellulose) Third session: Placebo patch and Placebo capsule (filler: methylcellulose)
Period: First Intervention (1 Day)
Arm/Group | Placebo, Nicotine, Mecamylamine | Nicotine, Placebo, Mecamylamine | Placebo, Mecamylamine, Nicotine | Nicotine, Mecamylamine, Placebo | Mecamylamine, Placebo, Nicotine | Mecamylamine, Nicotine, Placebo
Started | 4 | 3 | 4 | 5 | 2 | 3
Completed | 4 | 3 | 4 | 4 | 2 | 3
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Placebo, Nicotine, Mecamylamine | Nicotine, Placebo, Mecamylamine | Placebo, Mecamylamine, Nicotine | Nicotine, Mecamylamine, Placebo | Mecamylamine, Placebo, Nicotine | Mecamylamine, Nicotine, Placebo
Started | 4 | 3 | 4 | 4 | 2 | 3
Completed | 3 | 3 | 4 | 4 | 2 | 3
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (1 Day)
Arm/Group | Placebo, Nicotine, Mecamylamine | Nicotine, Placebo, Mecamylamine | Placebo, Mecamylamine, Nicotine | Nicotine, Mecamylamine, Placebo | Mecamylamine, Placebo, Nicotine | Mecamylamine, Nicotine, Placebo
Started | 3 | 3 | 4 | 4 | 2 | 3
Completed | 3 | 3 | 4 | 3 | 2 | 3
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Non-compliance (slept) | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 21 healthy non-smokers were randomized.
Groups:
- All Study Participants: Participants in each of the six arms received all three interventions (placebo, nicotine, mecamylamine).
Arm/Group | All Study Participants
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Reaction Time
Description: average reaction time on cognitive task performed in the MR scanner
Time Frame: 1 day
Population: 18 healthy male and female adult non-smokers. Only study completers are included, due to the within-subject design.
Measure: Mean (95% Confidence Interval); unit: ms
Groups:
- Intervention: Placebo: A placebo patch and a placebo capsule are administered.
- Intervention: Nicotine: A nicotine patch and a placebo capsule is administered.
- Intervention: Mecamylamine: A placebo patch and a mecamylamine capsule are administered.
Arm/Group | Intervention: Placebo | Intervention: Nicotine | Intervention: Mecamylamine
Number analyzed (Participants) | 18 | 18 | 18
ms
  Attention task reaction time | 512 [485 to 539] | 492 [464 to 520] | 524 [489 to 559]
  Working memory task reaction time | 541 [516 to 566] | 533 [508 to 558] | 573 [537 to 609]

2. Primary Outcome: Signal Detection Performance
Description: Signal detection on cognitive tasks performed in the MR scanner. For the attention task, this represents the percentage of trials in which the participant responded when a signal was presented. In the working memory task (N-back task), this represents the percentage of all target sequences to which the participant responded.
Time Frame: 1 day
Population: Healthy adult non-smokers (only study completers).
Measure: Mean (95% Confidence Interval); unit: percentage of all targets
Groups:
- Intervention: Nicotine: A nicotine patch and a placebo capsule are administered.
Arm/Group | Intervention: Placebo | Intervention: Nicotine | Intervention: Mecamylamine
Number analyzed (Participants) | 18 | 18 | 18
percentage of all targets
  Attention task correct identifications | 86.4 [81.4 to 91.4] | 93.8 [90.1 to 97.5] | 85.2 [79.7 to 90.7]
  Working memory task correct detections | 89.6 [88.4 to 90.8] | 95.5 [94.9 to 96.1] | 88.6 [87.9 to 89.3]

3. Primary Outcome: Default Network Activity
Description: Cognitive task-induced default network deactivation, measured by functional Magnetic Resonance Imaging. The default network was probed by five pre-defined ROIs per hemisphere. Task-induced deactivation was averaged across all ROIs.
Time Frame: 1 day
Population: Healthy non-smokers (only study completers).
Measure: Mean (95% Confidence Interval); unit: percentage of task-induced signal change
Groups:
- Intervention: Placebo: A placebo patch and a placebo capsule is administered.
Arm/Group | Intervention: Placebo | Intervention: Nicotine | Intervention: Mecamylamine
Number analyzed (Participants) | 18 | 18 | 18
percentage of task-induced signal change | -0.29 [-0.41 to -0.17] | -0.24 [-0.39 to -0.09] | -0.21 [-0.33 to -0.09]

4. Secondary Outcome: Subjective State
Description: End-of-session subjective state is measured by the Profile of Mood States (POMS). We utilize "Total Mood Disturbance" (TMD) as a summary measure, derived by adding the total scores on the five negative mood scales (tension, depression, anger, fatigue, confusion) and subtracting the score on the one positive mood scale (vigor). The theoretical range of the TMD scale is -32 to 228, with negative values indicating less mood disturbance, i.e., a more positive emotional state.
Time Frame: 1 day
Population: Healthy non-smokers (only study completers).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Intervention: Mecamylamine: A placebo patch and a mecamylamine capsule were administered.
Arm/Group | Intervention: Placebo | Intervention: Nicotine | Intervention: Mecamylamine
Number analyzed (Participants) | 18 | 18 | 18
units on a scale | -6.7 [-12.3 to -1.1] | -9.9 [-15.4 to -4.4] | -5.8 [-12 to 0.4]

5. Secondary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure (mmHg)
Time Frame: Bi-hourly: prior to patch application, 2 hours, 4 hours, and 6 hours after, and after the MRI scan (~8 hours after patch application)
Population: Healthy non-smokers
Measure: Mean (Standard Deviation); unit: mmHG
Groups:
- Intervention: Placebo: A placebo patch and a placebo capsule were administered.
- Intervention: Nicotine: A nicotine patch and a placebo capsule were administered.
Arm/Group | Intervention: Placebo | Intervention: Nicotine | Intervention: Mecamylamine
Number analyzed (Participants) | 18 | 18 | 18
mmHG
  Pre-patch | 120.2 (11.4) | 120.9 (16.7) | 119.3 (14.8)
  2 hours post patch | 116.1 (11.9) | 114.3 (10.7) | 112.3 (8.6)
  4 hours post patch | 120.1 (16.7) | 119.1 (9.9) | 114.4 (11.4)
  6 hours post patch | 120.3 (12.9) | 122.7 (12.7) | 118.2 (14.1)
  Post-scan | 129.7 (16.1) | 127.4 (9.8) | 121.5 (13.8)

6. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure in mmHg.
Time Frame: as for outcome 5
Population: Healthy non-smokers (only study completers).
Measure: Mean (Standard Deviation); unit: mmHG
Groups:
- Intervention: Placebo: Placebo patch and placebo capsule.
- Intervention: Nicotine: Nicotine patch and placebo capsule.
- Intervention: Mecamylamine: Placebo patch and mecamylamine capsule.
Arm/Group | Intervention: Placebo | Intervention: Nicotine | Intervention: Mecamylamine
Number analyzed (Participants) | 18 | 18 | 18
mmHG
  Pre-patch | 74.4 (8.0) | 71.6 (10.0) | 73.4 (10.1)
  2 hours post patch | 73.4 (10.0) | 71.9 (9.9) | 73.2 (9.7)
  4 hours post patch | 73.7 (9.7) | 71.1 (7.9) | 72.4 (6.9)
  6 hours post patch | 75.8 (6.6) | 75.3 (5.8) | 75.2 (8.1)
  Post-scan | 81.3 (5.4) | 81.1 (5.7) | 79.6 (9.4)

ADVERSE EVENTS:
Time Frame: 1 day (on each of separate 3 test days)
Groups:
- Intervention: Placebo: Participants receive a placebo patch and a placebo capsule.
- Intervention: Nicotine: Participants receive a nicotine patch and a placebo capsule.
- Intervention: Mecamylamine: Participants receive a placebo patch and a mecamylamine capsule.
Arm/Group | Intervention: Placebo | Intervention: Nicotine | Intervention: Mecamylamine
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 0/20 | 2/21 | 0/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention: Placebo (N=20) | Intervention: Nicotine (N=21) | Intervention: Mecamylamine (N=19)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No